CLINICAL TRIAL: NCT05065970
Title: A Double Blind, Randomized, Placebo-Controlled, Multicenter Phase IIa, Clinical Trial to Assess Efficacy and Safety of the Human Anti-CD38 Antibody Felzartamab in IgA Nephropathy
Brief Title: Clinical Trial to Assess Efficacy and Safety of the Human Anti-CD38 Antibody Felzartamab (MOR202) in IgA Nephropathy
Acronym: IGNAZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HI-Bio, A Biogen Company (Industry)
Responsible Party: Sponsor
Organization: Biogen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOR202C206
Record Dates: First submitted 2021-09-14; First posted 2021-10-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Immunoglobulin A (IgA) Nephropathy
Keywords: Kidney Disease; Urologic Disease; Glomerular Disease; Berger Disease; Glomerulonephritis, IGA
MeSH Terms: conditions — Kidney Diseases; Urologic Diseases; Glomerulonephritis, IGA | interventions — felzartamab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Felzartamab Arm #1 (Experimental)
  Interventions: Drug: Felzartamab
- Felzartamab Arm #2 (Experimental)
  Interventions: Drug: Felzartamab
- Felzartamab Arm #3 (Experimental)
  Interventions: Drug: Felzartamab

INTERVENTIONS:
Drug: Felzartamab — anti-CD38+ monoclonal antibody
  Other Names: MOR202
  Arms: Felzartamab Arm #1; Felzartamab Arm #2; Felzartamab Arm #3
Other: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled, multi-center, double-blind, proof of concept phase IIa trial and dose evaluation trial of felzartamab in IgAN

DETAILED DESCRIPTION:
Study Sponsor, originally HI-Bio, Inc., is now HI-Bio, A Biogen Company.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients ≥ 18 to ≤ 80 years (at date of signing the informed consent form [ICF]), but at least of legal age in the given country
* Biopsy confirmed diagnosis of IgAN within the past 8 years prior to signature of the ICF
* Proteinuria at screening visit ≥ 1.0 g/d.
* Treatment with an angiotensin-converting enzyme inhibitor (ACEi) and/or angiotensin receptor blocker (ARB) at maximum doses or maximally tolerated doses for ≥ 3 months prior to date of informed consent and adequate blood pressure (BP) control.
* A female of childbearing potential (FCBP), is only eligible to participate if she is not pregnant, not breast feeding, and agrees to follow the contraceptive guidance during the treatment period and for at least 3 months after the last dose of IMP

Key Exclusion Criteria:

* Hemoglobin < 90 g/L
* Thrombocytopenia: Platelets < 100.0 x 10^9/L.
* Neutropenia: Neutrophils < 1.5 x 10^9/L.
* Leukopenia: Leukocytes < 3.0 x 10^9/L
* Diabetes mellitus type 1
* Aspartate aminotransferase or alanine aminotransferase >1.5 x ULN, alkaline phosphatase >3.0 x ULN

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Efficacy: Relative change in Proteinuria value | 9 months compared to baseline

SECONDARY OUTCOMES:
Safety: determined by the frequency, incidence and severity of TEAEs | Ongoing through study completion, up to 2 years
Efficacy: Relative change in proteinuria value | Ongoing through treatment completion, an average every 3 months per treatment period, up to 2 years
Efficacy: complete response in patients with IgAN | Ongoing through treatment completion, an average every 3 months per treatment period, up to 2 years
Pharmacokinetic: serum concentrations of Felzartamab over time | Ongoing through treatment completion, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — HI-Bio, A Biogen Company
Locations (60):
- United States (4):
  - FOMAT Medical Research - FOMAT - HyperCore - PPDS, Oxnard, California
  - Amicis Research Center, Vacaville, Vacaville, California
  - Mayo Clinic Hospital - Methodist Campus, Rochester, Minnesota
  - MedResearch INC, El Paso, Texas
- Australia (2):
  - Core Research Group, Milton, Queensland
  - Sunshine Hospital - Australia, Saint Albans, Victoria
- Belgium (4):
  - Imelda VZW, Bonheiden, Antwerpen
  - UZ Leuven Hospital, Leuven, Vlaams Brabant
  - Regionaal Ziekenhuis Jan Yperman VZW, Ieper
  - CHU Sart Tilman Hospital, Liège
- Bulgaria (4):
  - Diagnostic- Consultative Center Convex EOOD, Sofia, Sofia-Grad
  - Medical Center Hera EOOD, Montana, Montana
  - Medical Center Hipokrat- N EOOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment, Stara Zagora
- Czechia (4):
  - Nemocnice AGEL Novy Jicin a.s, Nový Jicín, Moravskoslezský kraj
  - Eticka komise Fakultni nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Fakultni nemocnice Kralovske Vinohrady Hospital, Prague, Praha, Hlavní Mesto
  - Vseobecna Fakultni Nemocnice V Praze, Prague, Praha, Hlavní Mesto
- Georgia (3):
  - JSC Evex Hospitals, Tbilisi
  - L. Managadze National Center of Urology LTD, Tbilisi
  - Tbilisi State Medical University's and Ingorokva's University Clinic of High Medical Technologies, Tbilisi
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Japan (9):
  - National Hospital Organization Chibahigashi National Hospital, Chiba, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaidô
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu-Shi, Hukuoka
  - Kurume University Hospital, Kurume-Shi, Hukuoka
  - Fukushima Medical University Hospital, Fukushima, Hukusima
  - JCHO Sendai Hospital, Sendai, Miyagi
  - Japanese Red Cross Ashikaga Hospital, Ashikaga-Shi, Tochigi
  - Juntendo University Hospital, Bunkyō-Ku, Tokyo
  - Osaka University Hospital, Suita-Shi, Ôsaka
- University Malaya Medical Centre, Pantai, Malaysia
- St Frances Cabrini Medical Center and Cancer Institute, Santo Tomas, Batangas, Philippines
- Serbia (5):
  - Clinical Centre of Vojvodina, Novi Sad, Vojvodina
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Hospital Centar Zvezdara, Belgrade
  - General Hospital Krusevac, Kruševac
  - University Clinical Center Nis, Niš
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam, Gyeonggido
  - Ajou University Hospital, Suwon, Gyeonggido
  - Konkuk University Medical Center, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si
- Spain (8):
  - Fundacio Puigvert, Badalona
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Ruber Juan Bravo (Grupo Quironsalud), Madrid
- Taiwan (3):
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - Far Eastern Memorial Hospital, Taipei
- Ukraine (4):
  - Municipal Non-profit Enterprise Ternopil Regional Clinical Hospital of Ternopil Regional Council, Ternopil, Ternopil Oblast
  - Communal Nonprofit Enterprise "Kyiv City Center of Nephrology and Dialysis", Kyiv
  - State Institution Institute of Nephrology of NAMS of Ukraine, Kyiv
  - Municipal Nonprofit Enterprise Zaporizhzhia Regional Clinical Hospital Zaporizhzhia Regional Council, Zaporizhzhia
- Kings College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Floege J, Lafayette R, Barratt J, Schwartz B, Manser PT, Patel UD, Shah M, Kivman L, Faulhaber N, Kraft T, Thakur A, Hartle S, Barbour SJ. Randomized, double-blind, placebo-controlled phase 2a study assessing the efficacy and safety of felzartamab for IgA nephropathy. Kidney Int. 2025 Oct;108(4):695-706. doi: 10.1016/j.kint.2025.05.028. Epub 2025 Jun 26. PMID 40581166
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] El Karoui K, Fervenza FC, De Vriese AS. Treatment of IgA Nephropathy: A Rapidly Evolving Field. J Am Soc Nephrol. 2024 Jan 1;35(1):103-116. doi: 10.1681/ASN.0000000000000242. Epub 2023 Sep 29. PMID 37772889